CLINICAL TRIAL: NCT06177223
Title: Cognitive Behavioural Therapy for Post-Traumatic Stress Disorder (PTSD) Among Women Victims of Domestic Violence in Shelter Homes: A Randomized Control Trial
Brief Title: Cognitive Behavioral Therapy for Post-Traumatic Stress Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Government College University Faisalabad (Other)
Responsible Party: Principal Investigator, Qasir Abbas, Dr. Qasir Abbas Assistant Professor Clinical Psychology, Government College University Faisalabad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: nazishghafoor14@gmail.com
Record Dates: First submitted 2023-12-05; First posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Cognitive Behavioral Therapy
Keywords: Cognitive Behavioral Therapy, Domestic Violence
MeSH Terms: interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Randomized control trial design would be used in this study. it would be two arm study and there would be two groups an experimental and wait-list control group. Experimental group will receive intervention and another group would be placed in waitlist. In this research , parallel group design would be used. We will give treatment to all participants in a parallel way. Allocation ratio and framework would be equivalence i.e., treatment group and control group would be equal number of participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Cognitive Behavioral Therapy based sessions would be conducted with women victims of domestic violence in shelter homes
  Interventions: Behavioral: Cognitive Behavioral therapy
- Waitlist Control Group (No Intervention): no intervention would be given to the participants

INTERVENTIONS:
Behavioral: Cognitive Behavioral therapy — CBT-based treatment plan would be designed to address PTSD and associated problems.
  Arms: Treatment Group

SUMMARY:
The current study is designed to measure the role of cognitive behavior therapy with PTSD patients. There are following objectives of this current study, such as

1. To examine the efficacy of CBT to overcome the severity level of PTSD and associated psychiatric problems.
2. To change negative thought patterns and dysfunctional cognition into functional thoughts and beliefs.
3. To build up social support, enhance the quality of life and refine mental health among patients with PTSD.
4. To check outs the association of PTSD with depression, intimate partner violence stigma, marital adjustment, and abuse.
5. This study would examine the efficacy of CBT to treat the severity of PTSD and associated problems (i.e. depressive symptoms, adjustment problems & discrimination) among women victims of domestic violence in shelter homes

DETAILED DESCRIPTION:
Participants

Participants would be recruited from different women's shelters Homes. An Initial sample would be included total 200 participants. The final sample would be comprise 60 participants with age ranges will be 20 to 60 years. For collecting the sample, the Simple Random Sampling technique would be used. In this research, women with PTSD would be divided into two equal groups that would be n= 30 as the control group and n=30 experimental group through random assignment (See Fig.1: CONSORT Flowchart Diagram). One group diagnosed with PTSD would be providing 10 to 12 sessions of CBT. One other group diagnosed with PTSD depending on n=30 would not be provided CBT sessions. This research will be divided into 3 parts. In first initial procedure will be performed in which participants will be selected by simple random sampling. All women who live in shelters will be part of the study. After choosing the participant demographic form will be filled out. In demographic form information related to participants will be taken. This information will consist of age, gender, marital status, sibling, children, education, and financial status. In the second step, a standardized tool will be used to measure the symptoms of post-traumatic stress disorder. The pre-test will be taken from participants following: 1) LWMAT will measure the marital adjustment level of participants, 2) IPVSS will be for assess partner violence stigma symptoms, Domestic Violence Scale to measure domestic violence, PHQ-9 for measuring depression level, and PCL-5 for PTSD related symptoms according to DSM 5TR. A participant who has a high rate of PCL-5 and shows PTSD symptoms will be chosen for the experiment. Further, participants will be divided into two groups. One group is the experimental group n=30 and the second will be the control group n=30. In the next step, CBT techniques will be provided to the experimental group by the trained therapist. Following CBT techniques will be provided psycho-education, behavioral activation, problem-solving, cognitive conceptualization, stigma reduction, and relapse prevention. Furthermore, the control group will not be provided with CBT techniques. At the end of this procedure, patients will be re-assessed through the same measures as the post-test. All these assessments will be interpreted according to a given method by the author. A paired t-test will be used to find a correlation between the pre-test and post-test. Statistics will be applied using SPSS 26.0. Session frequency will be once a week and last approximately 40-45 minutes. The tentative duration would be 3 months. The session would be conducted one-on-one sitting in the women's shelter setting.

Eligibility Criteria

Participants that will be participated in this research would be Women who experienced domestic violence and who are meeting the DSM-V diagnostic criteria of PTSD with at least one year of history of marital issues. Only those women who live in the Shelters will be part of the research. Women with separation, divorced/widowed, single, and with medical comorbidity will be excluded from the study. Women who have physical problems will be excluded. Those women who intended to research will be part of the research. Women who have no PTSD symptoms will be excluded. The age ranges between 20 to 50 years will be included. Greater than 50 years and less than 20 years women will be excluded.

Interventions

CBT-based treatment plan would be designed to address PTSD and associated problems. 10-12 sessions will be structured having particular agendas. In each session, the therapist would try to achieve the target goal using particular techniques, interventions, and modalities to address the target goals.

Expected outcomes

CBT will treat cognitive distortions, negative feelings and emotions, and irrational beliefs, which are associated with trauma as well as improve social interaction, trauma reduction, marital satisfaction, and daily life functioning.

ELIGIBILITY:
Inclusion Criteria:

* Women who experienced domestic violence
* Diagnosed women of PTSD from DSM-V
* Women with at least one year of history of marital issues
* Women living in the Shelters
* Intended to Research

Exclusion Criteria:

* Divorced/widowed, Single
* Women with medical comorbidity
* Women with physical problems
* Minimum to 20 years of age
* Maximum to 50 years

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — only married women and those who are living in shelter home would be part of the study
Enrollment: 200 (Estimated)
Dates: Start 2023-11-10 (Actual); Primary Completion 2024-01-30 (Estimated); Study Completion 2024-04-10 (Estimated)

PRIMARY OUTCOMES:
Post Traumatic Stress Disorder | 3-5 weeks
  The Post Traumatic Stress Disorder assessed by PTSD Checklist for Diagnostic and Statistical Manual of Mental Health Disorder-Fifth Edition (PCL-5) is a 20-item self-report measure. A total symptom severity score (range _0-80) can be obtained by summing the scores for each of the 20 items. Cutoff score between 31-33 indicative diagnosis of PTSD.
Domestic Violence | after allocation (1 week)
  Karachi domestic violence screening scale used to measure intimate partner violence. It contains 35 items having 5 subscales i.e., physical abuse, psychological abuse, sexual abuse, victim characteristic, abuser characteristic. Total score ranges between 0 to 105 and cut off score is 30. Score ranges categorized as no abuse= 0-19, mild= 20-35, moderate= 36-59, severe= 60-105.
Depression | after allocation (1 week)
  Depression will be assessed by using Patient Health Questionnaire-9. The total scores of 5, 10, 15, and 20 are taken as mild, moderate, moderately severe, and severe respectively.
Marital Adjustment | after allocation (1 week)
  Locke Wallace Marital Adjustment Test used to measure adjustment level in married couples as high or low and agreement or disagreement on the cause of conflicted issues as well. It's score ranges from 2 to 158. The cut off score is 100, which indicate maladjustment in marital life. High score reflects high rate of satisfaction.
Intimate partner Violence Stigma | after allocation (1 week)
  The intimate partner violence stigma scale used for measuring stigma associated to intimate partner violence. This scale has four subscales that measure stigma including anticipated stigma, perpetrator stigma, internalized stigma, and isolation. High score indicate high stiga.

CONTACTS AND LOCATIONS:
Overall Officials: Qasir Abbas, PHD, Principal Investigator — Government College University, Faislabad.
Locations (1):
- Dr. Qasir Abbas, Faisalabad, Province, Pakistan

IPD SHARING:
Plan to Share IPD: No